CLINICAL TRIAL: NCT04846101
Title: Evaluation of Shade Matching Capacity of a Single-shade Contemporary Resin Composite in Anterior Restorations
Brief Title: Evaluation of Shade Matching Capacity of a Contemporary Composite Dental Material
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of Trial components
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Susan Hattar, Associate Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCTomnishade
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Dental Restoration
Keywords: shade matching, dental material, blending effect

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blind Observers will be asked to assess the shade matching capacity of the restorative material on a Likert Scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior restorations using single shade OMNICHROMA composite (Experimental): Anterior class III and Class IV cavities will be restored using single shade composite material according to standard protocols of etching, bonding and composite placement.
  Interventions: Other: OMNISHADE; Diagnostic Test: Instrumental Shade Analysis; Other: Visual Shade Analysis; Other: Patient satisfaction
- Anterior restorations using multi-shade composite (Active Comparator): Shade selection for the tooth will be performed prior to the placement of the restoration. Anterior class III and Class IV cavities will be restored using multi-shade composite material according to standard protocols of etching, bonding and composite placement.
  Interventions: Other: MULTISHADE; Diagnostic Test: Instrumental Shade Analysis; Other: Visual Shade Analysis; Other: Patient satisfaction

INTERVENTIONS:
Other: OMNISHADE — Anterior dental cavities (Class III, Class IV) will be restored with an omnishade composite material
  Arms: Anterior restorations using single shade OMNICHROMA composite
Other: MULTISHADE — Anterior dental cavities (Class III, Class IV) will be restored with conventional multishade composite material.
  Arms: Anterior restorations using multi-shade composite
Diagnostic Test: Instrumental Shade Analysis — Assessment will be performed by single operator using spectrophotometer (EASYSHADE) to detect color difference between tooth and restoration
Other: Visual Shade Analysis — Visual assessment will be performed by two calibrated specialists to evaluate shade matching between the tooth and restoration
Other: Patient satisfaction — Patient satisfaction of the final shade match will be assessed on a visual analogue scale

SUMMARY:
One of the main difficulties encountered in esthetic dentistry is the complexity associated with shade matching and layering technique to achieve optimal esthetic outcomes. To ensure an esthetic outcome, an imperceptible match of the color of the restorative material to that of the tooth is of utmost importance. Recently, a new shade matching composite that utilizes "smart chromatic technology", developed by Tokuyama was claimed to be able to capture the structural color of its surroundings teeth. Our main objective is to assess the blending capacity of OMNICHROMA composite material in anterior restorations of patients attending the Jordan University Hospital. Both visual and instrumental measurements will be performed and the differences between the shade of the composite resin and the tooth structure will be measured. In addition, multi chroma composite restorations will be placed for the purpose of comparison (control).

DETAILED DESCRIPTION:
In the present study, the restorations will be placed under rubber dam isolation for moisture control. The cavities will be prepared according to the concepts of minimal invasive dentistry. Prior to placing the composite resin, the margins of the cavities will be finished using ultra fine grit diamond burs·and beveled in a 1-mm area. Deep cavities suspected to be near the pulp be lined with RMGI. Inclusion criteria: class Ill and Class IV carious lesions.

The enamel margins of the cavities will be acid etched for 60s with 37% phosphoric acid and then rinsed thoroughly with water spray. Afterwards, the dentin bonding system will be applied, left undisturbed for 20 s and then excess removed using an air syringe and light cured for 20s. The restorative composite material will be placed in incremental layers, adapted, each layer cured for 40s. After polymerization, the restorations will be finished under profuse water spray using diamonds, Sof-Lex finishing discs and polishers.

All restorations will be placed by one dentist (Pl). Written informed consent will be provided to all participants prior to starting the treatment

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients
* Patients requiring anterior restorations
* Vital teeth
* Absence of periodontal or pulpal disease
* Patients willing to sign informed consent and returning for follow up

Exclusion Criteria:

* Patients with extensive caries and tooth loss
* Patient with periodontal disease
* Patients with poor oral hygiene and lack of motivation
* Patient with severe extrinsic or intrinsic discolorations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Instrumental Color assessment | 2 years
  Color difference between restoration & tooth will be assessed using VITASHADE spectrophotometer
Visual color assessment | 2 years
  Color difference between restoration & tooth will be evaluated by independent observers

SECONDARY OUTCOMES:
Patient satisfaction | 2 years
  Patient satisfaction of shade matching of the restoration will be evaluated using visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- The university ofJordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available for other researchers
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 2 years

REFERENCES:
- [Background] Mikhail SS, Schricker SR, Azer SS, Brantley WA, Johnston WM. Optical characteristics of contemporary dental composite resin materials. J Dent. 2013 Sep;41(9):771-8. doi: 10.1016/j.jdent.2013.07.001. Epub 2013 Jul 12. PMID 23851132
- [Background] Paravina RD, Westland S, Kimura M, Powers JM, Imai FH. Color interaction of dental materials: blending effect of layered composites. Dent Mater. 2006 Oct;22(10):903-8. doi: 10.1016/j.dental.2005.11.018. Epub 2005 Dec 27. PMID 16378637
- [Background] Paravina RD, Westland S, Imai FH, Kimura M, Powers JM. Evaluation of blending effect of composites related to restoration size. Dent Mater. 2006 Apr;22(4):299-307. doi: 10.1016/j.dental.2005.04.022. Epub 2005 Aug 8. PMID 16085303
- [Background] Tanaka A, Nakajima M, Seki N, Foxton RM, Tagami J. The effect of tooth age on colour adjustment potential of resin composite restorations. J Dent. 2015 Feb;43(2):253-60. doi: 10.1016/j.jdent.2014.09.007. Epub 2014 Sep 19. PMID 25242100
- [Background] Pereira Sanchez N, Powers JM, Paravina RD. Instrumental and visual evaluation of the color adjustment potential of resin composites. J Esthet Restor Dent. 2019 Sep;31(5):465-470. doi: 10.1111/jerd.12488. Epub 2019 May 16. PMID 31095870